CLINICAL TRIAL: NCT04754126
Title: Amazing Me: A Body Confidence Health and Wellness Program for 4th and 5th Graders
Brief Title: Efficacy Study of Amazing Me Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Marisol Perez, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00012339
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Self Esteem; Body Distorted Images
Keywords: body satisfaction; self esteem; weight-based bullying and teasing

STUDY DESIGN:
Intervention Model Description: A randomized controlled trail will be conducted to ascertain the effectiveness of the Amazing Me intervention in 9-11 year old children. The randomized controlled trial will consist of an intervention and control group. Between 100 to 180 classrooms will be randomized to control or intervention condition. Randomization distribution will be 50%; thus, half of the educators/classrooms will be in the intervention and half in the control. We estimate about 30 students per teacher, yielding a maximum of 2,700 students randomized to intervention and 2,700 students randomized to control. Educators and school districts will be recruited to participate. Educators and students will complete an online baseline survey and another survey after the intervention. Finally, a 6-month and 12-month follow-up survey will be conducted for students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Educators and students complete a baseline survey. Educators will implement 6 lessons, each 45 minutes, in the classroom. Educators are free to choose the time between lessons, so some can implement all in one week, others can choose to implement once per week. Educators are given a maximum of 6 weeks to implement the curriculum. Educators and students complete a post-program survey. Students complete a 6- and 12-month follow-up survey.
  Interventions: Behavioral: Amazing Me
- Control Group (No Intervention): This group will only complete online surveys that match the time when intervention group is complete the surveys. There is a baseline survey and then a post-survey 6 weeks later for both educators and students. Additionally, students will complete a 6- and 12-month follow-up survey.

INTERVENTIONS:
Behavioral: Amazing Me — The Amazing Me Program is an evidence-based program designed to help children between the ages of 9 and 11 build self-esteem, body confidence, and eliminate weight-based bullying and teasing. This school-based curriculum satisfies national educational health requirements and provides tools for teachers to implement in 4th and 5th grade classrooms.
  Arms: Intervention Group

SUMMARY:
The objective of the Efficacy Study of Amazing Me Program is to deliver the Amazing Me intervention and assess its efficacy. The Amazing Me intervention aims to help children between the ages of 9 and 11 build self-esteem, body confidence, and eliminate weight-based bullying and teasing. The Amazing Me intervention teaches students to be kind to themselves, their bodies, and to others.

DETAILED DESCRIPTION:
Body dissatisfaction is one of the most robust risk factors for developing unhealthy behaviors, low self-esteem, and contributes to anxiety and depression in adolescence. Despite evidence that body dissatisfaction can emerge during the elementary school years, the majority of body confidence programs are for girls over the age of 15. There is very little to no research on interventions for elementary school children. The Body Project is an empirically supported body confidence prevention program for high school girls with over 100 articles to support its efficacy, effectiveness and theoretical model; it is the only body confidence program for youth to acquire the Blueprints Certification. Together with two 4th and 5th grade teachers, the investigators have adapted the Body Project curriculum for youth between the ages of 9 to 11 years old (i.e., 4th and 5th graders). The curriculum is called Amazing Me and will be implemented in classrooms by teachers. The curriculum was developed meeting several competencies for national health and wellness standards for elementary students. The aim of the current study is to conduct a national randomized control trial of the curriculum 100 classrooms with 4th and 5th graders.

The primary aim of the current study is to deliver the Amazing Me intervention and assess its efficacy. It is hypothesized that compared to controls, children that undergo the body confidence curriculum will report higher body satisfaction and body esteem scores, overall greater self-esteem, and will report less engagement in appearance comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Educators teaching 4th and 5th graders. Thus students will be on average between 9 and 11 years old.

Exclusion Criteria:

* None.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Body-Esteem Scale | Baseline,
  The Body-Esteem Scale is a 24-item self-report measure designed for use with children. The items were developed to assess how children feel about themselves and how they believe others view them. Sample items include "I like what I look like in pictures" and "There are lots of things I'd change about my looks if I could." Children responded by selecting "yes" or "no" for each item. In this study, children were also given the option of selecting "I don't want to answer." This scale has been found to be a reliable measure of body esteem in children as young as 7 years old. All items from this scale were used in the pilot study.
Body-Esteem Scale | 6 weeks after baseline
  The Body-Esteem Scale is a 24-item self-report measure designed for use with children. The items were developed to assess how children feel about themselves and how they believe others view them. Sample items include "I like what I look like in pictures" and "There are lots of things I'd change about my looks if I could." Children responded by selecting "yes" or "no" for each item. In this study, children were also given the option of selecting "I don't want to answer." This scale has been found to be a reliable measure of body esteem in children as young as 7 years old. All items from this scale were used in the pilot study.
Body-Esteem Scale | 9-12 month follow up
  The Body-Esteem Scale is a 24-item self-report measure designed for use with children. The items were developed to assess how children feel about themselves and how they believe others view them. Sample items include "I like what I look like in pictures" and "There are lots of things I'd change about my looks if I could." Children responded by selecting "yes" or "no" for each item. In this study, children were also given the option of selecting "I don't want to answer." This scale has been found to be a reliable measure of body esteem in children as young as 7 years old. All items from this scale were used in the pilot study.
Physical Appearance Related Teasing Scale | Baseline
  The Physical Appearance Related Teasing Scale was adapted for the current study. The original scale consists of 18 items with two factors: weight/size teasing and general appearance teasing. Items 1, 2, 3, 4, 5, 6, 14, 16, 17, 18 were used in the current study. Items 1-6 load onto the weight/size teasing factor and items 14, 16, 17-18 load onto the general appearance teasing factor. Items were modified to be developmentally appropriate. The Perception of Teasing Scale (POTS) was incorporated to measure perceptions of distress where participants were asked to rate the degree to which they were upset by the teasing on a 3-point Likert scale ranging from 1 (not upset) to 3 (very upset), modified from the original The POTS was originally developed with adults and has been used extensively with children and adolescents.
Physical Appearance Related Teasing Scale | 6 weeks after baseline
  The Physical Appearance Related Teasing Scale was adapted for the current study. The original scale consists of 18 items with two factors: weight/size teasing and general appearance teasing. Items 1, 2, 3, 4, 5, 6, 14, 16, 17, 18 were used in the current study. Items 1-6 load onto the weight/size teasing factor and items 14, 16, 17-18 load onto the general appearance teasing factor. Items were modified to be developmentally appropriate. The Perception of Teasing Scale (POTS) was incorporated to measure perceptions of distress where participants were asked to rate the degree to which they were upset by the teasing on a 3-point Likert scale ranging from 1 (not upset) to 3 (very upset), modified from the original The POTS was originally developed with adults and has been used extensively with children and adolescents.
Physical Appearance Related Teasing Scale | 9-12 month follow up
  The Physical Appearance Related Teasing Scale was adapted for the current study. The original scale consists of 18 items with two factors: weight/size teasing and general appearance teasing. Items 1, 2, 3, 4, 5, 6, 14, 16, 17, 18 were used in the current study. Items 1-6 load onto the weight/size teasing factor and items 14, 16, 17-18 load onto the general appearance teasing factor. Items were modified to be developmentally appropriate. The Perception of Teasing Scale (POTS) was incorporated to measure perceptions of distress where participants were asked to rate the degree to which they were upset by the teasing on a 3-point Likert scale ranging from 1 (not upset) to 3 (very upset), modified from the original The POTS was originally developed with adults and has been used extensively with children and adolescents.
Rosenberg Self-Esteem Scale | Baseline
  A 10-item scale that measures global self-esteem by measuring both positive and negative feelings about the self. Items were modified to be developmentally appropriate for children. Example items include "I like myself" and "I feel there are a lot of good things about me." The scale is uni-dimensional. All items are answered using a 4-point Likert scale format ranging from "strongly agree" to "strongly disagree." In this study, children were also given the option of selecting "I don't want to answer." All items from this scale were used in the pilot study.
Rosenberg Self-Esteem Scale | 6 weeks after baseline
  A 10-item scale that measures global self-esteem by measuring both positive and negative feelings about the self. Items were modified to be developmentally appropriate for children. Example items include "I like myself" and "I feel there are a lot of good things about me." The scale is uni-dimensional. All items are answered using a 4-point Likert scale format ranging from "strongly agree" to "strongly disagree." In this study, children were also given the option of selecting "I don't want to answer." All items from this scale were used in the pilot study.
Rosenberg Self-Esteem Scale | 9-12 month follow up
  A 10-item scale that measures global self-esteem by measuring both positive and negative feelings about the self. Items were modified to be developmentally appropriate for children. Example items include "I like myself" and "I feel there are a lot of good things about me." The scale is uni-dimensional. All items are answered using a 4-point Likert scale format ranging from "strongly agree" to "strongly disagree." In this study, children were also given the option of selecting "I don't want to answer." All items from this scale were used in the pilot study.

SECONDARY OUTCOMES:
Teacher Satisfaction Scale | baseline
  This is a three item measure assessing satisfaction with curriculum, on a 5-point Likert scale.
Teacher Satisfaction Scale | 6 weeks after baseline
  This is a three item measure assessing satisfaction with curriculum, on a 5-point Likert scale.
Fidelity and Adherence Coding | 6 weeks after baseline
  This is a 10 item measure coded by raters assessing the extent to which teacher's administer the program as prescribed
Knowledge Check Test | baseline
  This is an 8 item measures that assesses comprehension and knowledge of the curriculum materials, concepts and goals
Knowledge Check Test | 6 weeks after baseline
  This is an 8 item measures that assesses comprehension and knowledge of the curriculum materials, concepts and goals
Knowledge Check Test | 9-12 month follow up
  This is an 8 item measures that assesses comprehension and knowledge of the curriculum materials, concepts and goals
Appearance Conversations Scale | baseline
  The Appearance Conversations Scale assesses the frequency with which participants report talking about their bodies and appearance with friends. In the original measure, responses are rated on a 5-point Likert scale ranging from "never" (1) to "very often" (5). In the current study, the scale was modified to a 3-point Likert scale ranging from "never" (1) to "a lot" (3) to be developmentally appropriate.
Appearance Conversations Scale | 6 weeks after baseline
  The Appearance Conversations Scale assesses the frequency with which participants report talking about their bodies and appearance with friends. In the original measure, responses are rated on a 5-point Likert scale ranging from "never" (1) to "very often" (5). In the current study, the scale was modified to a 3-point Likert scale ranging from "never" (1) to "a lot" (3) to be developmentally appropriate.
Appearance Conversations Scale | 9-12 month follow up
  The Appearance Conversations Scale assesses the frequency with which participants report talking about their bodies and appearance with friends. In the original measure, responses are rated on a 5-point Likert scale ranging from "never" (1) to "very often" (5). In the current study, the scale was modified to a 3-point Likert scale ranging from "never" (1) to "a lot" (3) to be developmentally appropriate.
Figure Rating Scale | baseline
  were developed based on adult figure drawings by Stunkard, Sorenson, and Schulsinger (1983). Figures were created to illustrate body weight ranging from very thin to obese. This scale can be used to assess preferences and perceptions of self, ideal self, ideal other child, other adult, and ideal other adult. In the current study, "self" and "other-gender" were used. For example, if participants identified as girls, they were presented with corresponding figure drawings for "self" ("which picture looks the most like you?") and figure drawings of boys for "other-gender" ("which picture shows the way you think is best for girls/boys to look?")
Figure Rating Scale | 6 weeks after baseline
  were developed based on adult figure drawings by Stunkard, Sorenson, and Schulsinger (1983). Figures were created to illustrate body weight ranging from very thin to obese. This scale can be used to assess preferences and perceptions of self, ideal self, ideal other child, other adult, and ideal other adult. In the current study, "self" and "other-gender" were used. For example, if participants identified as girls, they were presented with corresponding figure drawings for "self" ("which picture looks the most like you?") and figure drawings of boys for "other-gender" ("which picture shows the way you think is best for girls/boys to look?")
Figure Rating Scale | 9-12 month follow up
  were developed based on adult figure drawings by Stunkard, Sorenson, and Schulsinger (1983). Figures were created to illustrate body weight ranging from very thin to obese. This scale can be used to assess preferences and perceptions of self, ideal self, ideal other child, other adult, and ideal other adult. In the current study, "self" and "other-gender" were used. For example, if participants identified as girls, they were presented with corresponding figure drawings for "self" ("which picture looks the most like you?") and figure drawings of boys for "other-gender" ("which picture shows the way you think is best for girls/boys to look?")

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Funder and IRB must first approve any sharing of IPD with other researchers.